CLINICAL TRIAL: NCT01869270
Title: Gene Therapy for Tay-Sachs Disease (Phase 1: Natural History Data Gather)
Brief Title: Gene Therapy for Tay-Sachs Disease
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0905M66723; U54NS065768 (NIH)
Record Dates: First submitted 2013-05-22; First posted 2013-06-05 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Tay Sachs Disease; Sandhoff Disease; Late Onset Tay Sachs Disease
Keywords: hexosaminidase deficiency; Tay-Sachs disease; Sandhoff disease; late-onset Tay-Sachs disease; adult-onset Tay-Sachs disease; late onset Tay Sachs disease; adult onset Tay Sachs disease; retrospective; hexosaminidase A activity; GM2-ganglioside; gangliosidoses; natural history; hexosaminidase
MeSH Terms: conditions — Tay-Sachs Disease; Sandhoff Disease; Gangliosidoses, GM2; Gangliosidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hypothesis: To study the natural history of Tay-Sachs disease and evaluate therapeutic interventions.

This study is intended to work in collaboration with NCT00668187 "A Natural History Study of Hexosaminidase Deficiency." Because so few patients with Tay-Sachs disease present annually, we will maximize both research projects by enrolling patients in both studies. For this present study, we will perform retrospective medical record review to gather data. Through this medical record review, we will collect biomarker analysis results, neuroimaging report data, quality-of-life questionnaire data and ophthalmology exam findings. If the subject has undergone therapy or treatment, the results will be noted.

DETAILED DESCRIPTION:
Much has been done in the past four decades to better understand, improve diagnostic measures of, and prevent hexosaminidase deficiency diseases, yet all of them - Tay-Sachs, Sandhoff, and Late Onset Tay-Sachs (LOTS) - remain diseases without treatment. Much work remains to be done to understand and effectively treat these diseases. To date, no comprehensive assessment of the natural history of Tay-Sachs or Sandhoff has been undertaken. The information that is gathered through this study will characterize and describe the Tay-Sachs disease population as a whole, including the variability and progression of this disease. This information, in turn, will function as a point of reference against which to assess the efficacy of therapeutic interventions. Therapeutic interventions may include any treatments/therapies the subject may have undergone in the past, including hematopoietic cell transplantation, and/or the administration of miglustat, acetylcysteine, or other pharmaceutical agents; and possible future gene therapies.

ELIGIBILITY:
Inclusion Criteria:

Any person who has been diagnosed with a hexosaminidase deficiency disease can be included in this study.

Exclusion Criteria:

The only exclusion criteria is a desire not to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any person, living or dead, who has been diagnosed with a hexosaminidase deficiency disease
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Biomarkers | Participants will be followed for the duration of the study, an expected average of two years.
  Biomarkers data to be collected include:
  1. CSF (cerebro-spinal fluid) hexosaminidase A activity
  2. CSF GM2-ganglioside
  3. CSF protein
  4. CSF chitotriosidase

SECONDARY OUTCOMES:
Results of Ancillary Therapies or Treatments | Participants will be followed for the duration of the study, an expected average of two years.
  The results of any ancillary therapies or treatments will be noted. Such therapies or treatments may include hematopoietic cell transplantation and/or pharmacologic interventions.
Clinical Indicators | Participants will be followed for the duration of the study, an expected average of two years.
  Clinical indicators data to be collected include:
  1. Cranial morphology from MRI exam reports
  2. Ophthalmologic exam findings
  3. Behavioral assessment and quality-of-life questionnaire responses from NCT00668187, which collaborates with the present study
  4. Life-span length

CONTACTS AND LOCATIONS:
Overall Officials: Chester B. Whitley, PhD, MD, Principal Investigator — University of Minnesota; Jeffrey Krischer, PhD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Data Management and Coordinating Center (DMCC), Univ. of South Florida, Tampa, Florida
  - University of Minnesota, Minneapolis, Minnesota